CLINICAL TRIAL: NCT03647761
Title: Does Wearing Tetra-Grip Improve Upper Extremity Function in Children Diagnosed With Neonatal Brachial Plexus Palsy?
Brief Title: Does Wearing Tetra-Grip Improve Arm Function in Children Diagnosed With Neonatal Brachial Plexus Palsy?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid19, lack of manpower
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Rinaldi, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 022018-069
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Neonatal Brachial Plexus Palsy
Keywords: Tetra-grip; Assisting Hand Assessment
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care
- Treatment (Experimental): Tetra-grip applied
  Interventions: Device: Tetra-grip

INTERVENTIONS:
Device: Tetra-grip — Tetra-grip is a tubular elastic bandage that provides both compression and support
  Arms: Treatment

SUMMARY:
This study evaluates the effect of wearing a tetra-grip on the affected arm of children with neonatal brachial plexus palsy. Half of the participants will have tetra-grip applied to the arm, while the other half will not have it applied to the arm.

DETAILED DESCRIPTION:
Tetra-grip is a tubular elastic support bandage that provides both compression and support. Previous studies have shown that by applying neoprene or athletic tape to a joint on individuals with poor proprioception or a history of joint injury, such modalities enhanced their proprioceptive recognition via stimulation of mechanoreceptors responding to skin stretch and compression during joint motion. As a result, patients have greater kinesthetic and joint position awareness of their limb.

ELIGIBILITY:
Inclusion Criteria:

* 3 - 7 years old
* male or female
* non-dominant upper extremity brachial plexus injury

Exclusion Criteria:

* Botox injections to the affected extremity within the past 3 months
* Severe muscle contractures of affected extremity that restricts functional use of the arm and hand
* Concurrent cerebral palsy

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | At the end of standard OT sessions usually lasting 3 months.
  AHA measures hand function evaluation for children with unilateral upper limb disabilities

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States